CLINICAL TRIAL: NCT06942234
Title: The Multicenter, Open-label, Single-arm, Multi-cohort Phase Ib/II Clinical Study to Evaluate the Efficacy and Safety of JSKN016 in Combination Therapy in Chinese Participants With Inoperable Locally Advanced or Metastatic HER2-negative Breast Cancer
Brief Title: Study of JSKN016 Combination Therapy in Inoperable Locally Advanced or Metastatic HER2-Negative Breast Cancer
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Jiangsu Alphamab Biopharmaceuticals Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JSKN016-202
Record Dates: First submitted 2025-04-10; First posted 2025-04-24 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Inoperable Locally Advanced HER2-Negative Breast Cancer; Metastatic HER2-Negative Breast Cancer
MeSH Terms: interventions — Capecitabine; Taxes; eribulin; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Cohort 1: JSKN016+Paclitaxel (Experimental): JSKN016 (5mg/kg IV Q3W D1) + nab-paclitaxel (125mg/m² IV Q3W D1, D8)
  Interventions: Drug: JSKN016; Drug: Paclitaxel (albumin bound)
- Cohort 2: JSKN016+Capecitabine (Experimental): JSKN016 (5mg/kg IV Q3W D1) + capecitabine (1000mg/m² PO BID Q3W D1-14)
  Interventions: Drug: JSKN016; Drug: Capecitabine
- Cohort 3: JSKN016+Eribulin (Experimental): JSKN016 (5mg/kg IV Q3W D1) + eribulin (1.4mg/m² IV Q3W D1, D8)
  Interventions: Drug: JSKN016; Drug: Eribulin
- Cohort 4: JSKN016+Pembrolizumab/Toripalimab (Experimental): JSKN016 (5mg/kg IV Q3W D1) + pembrolizumab (200mg IV Q3W D1) or toripalimab (240mg IV Q3W D1).
  Interventions: Drug: JSKN016; Drug: Pembrolizumab

INTERVENTIONS:
Drug: JSKN016 — JSKN016 is administered via intravenous infusion at doses of 5mg/kg or 6mg/kg every 3 weeks, starting on Day 1 of each cycle. If the 5mg/kg dose is well tolerated during the safety lead-in phase, the dose may be increased to 6mg/kg for subsequent cycles.
Drug: Capecitabine — The drug is administered orally at a dose of 1000mg/m², twice daily for two weeks, followed by a one-week break. Treatment cycles repeat every three weeks.
  Arms: Cohort 2: JSKN016+Capecitabine
Drug: Paclitaxel (albumin bound) — The drug is administered intravenously at a dose of 125mg/m², with infusions on Day 1 and Day 8 of each treatment cycle. The treatment cycle is repeated every 3 weeks.
  Arms: Cohort 1: JSKN016+Paclitaxel
Drug: Eribulin — The drug is administered intravenously at a dose of 1.4mg/m², with infusions on Day 1 and Day 8 of each treatment cycle. The treatment cycle is repeated every 3 weeks.
  Arms: Cohort 3: JSKN016+Eribulin
Drug: Pembrolizumab — The drug is administered intravenously at a fixed dose of 200mg, with infusions on Day 1 of each 3-week treatment cycle.
  Arms: Cohort 4: JSKN016+Pembrolizumab/Toripalimab

SUMMARY:
This study aims to evaluate the safety and effectiveness of JSKN016 in combination with different treatments for patients with HER2-negative breast cancer that cannot be removed by surgery or has spread to other parts of the body. The study includes four groups of patients based on treatment history and tumor characteristics. Each group will receive JSKN016 with chemotherapy or immunotherapy. The goal is to find out how well the treatment works and how safe it is.

DETAILED DESCRIPTION:
This clinical study investigates the safety and efficacy of JSKN016 combined with various therapies for patients with advanced, inoperable, or metastatic HER2-negative breast cancer. The study includes four groups with different treatment regimens, targeting HR+HER2-negative breast cancer and triple-negative breast cancer (TNBC) with varying prior treatments. Participants will receive JSKN016 in combination with paclitaxel, capecitabine, eribulin, or pembrolizumab. The primary endpoint is the objective response rate (ORR) based on RECIST 1.1 criteria. The secondary endpoints include efficacy, safet, and other related outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Capable of understanding and signing the informed consent form.
2. Aged ≥18 and ≤75 years, regardless of sex.
3. Histologically or cytologically confirmed inoperable locally advanced or metastatic HER2-negative breast cancer.
4. Hormone receptor-positive participants with progression/intolerance after standard endocrine therapy, or unsuitable for it.
5. Disease progression confirmed by radiological evidence post-systemic treatment.
6. Available archived or newly obtained tumor tissue/biopsy.
7. No prior systemic therapy for advanced disease, except for prior endocrine ± targeted therapy or CDK4/6 inhibitors.
8. Measurable non-CNS lesion per RECIST 1.1.
9. Expected survival ≥3 months.
10. ECOG performance status of 0 or 1.
11. Contraceptive use agreement for fertile participants.
12. Adequate organ function within 7 days of enrollment:

    * Bone marrow: ANC ≥1.5 × 10⁹/L, Hemoglobin ≥90 g/L, Platelets ≥100 × 10⁹/L.
    * Liver: Bilirubin ≤1.5 × ULN, ALT/AST ≤3 × ULN.
    * Renal: Creatinine ≤1.5 × ULN or Ccr ≥60 mL/min.
    * Coagulation: INR/PT ≤1.5 × ULN, APTT ≤1.5 × ULN.
13. LVEF ≥50%.

Exclusion Criteria:

1. CNS metastasis (except stable cases treated with radiation or surgery).
2. Unstable spinal cord compression or untreated history.
3. Recent live vaccine (except seasonal flu vaccines).
4. Recent anti-tumor treatment within 28 days or 5 half-lives (whichever is shorter).
5. Recent palliative therapy within 14 days.
6. Major surgery within 28 days or planned during the study.
7. Severe gastrointestinal issues or recent major GI bleeding.
8. Uncontrolled pleural/peritoneal effusions or cachexia.
9. Prior HER3/TROP2-targeted therapy or topoisomerase I inhibitors.
10. Other malignancies within 5 years (except certain skin or localized cancers).
11. Current interstitial lung disease or uncontrolled infections.
12. Severe hypercalcemia or uncontrolled cancer-related pain.
13. Autoimmune diseases, unless stable with treatment.
14. Uncontrolled comorbidities (e.g., active infections, cardiovascular issues).
15. Toxicities from previous treatments not resolved to CTCAE ≤1.
16. Recent steroid use or need for systemic immunosuppressive therapy.
17. Allergy to study drug components.
18. Pregnancy or breastfeeding.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Objetctive Response Rate (ORR) | From baseline until disease progression, death, or end of treatment, whichever occurs first (up to approximately 24 months)
  The proportion of participants who achieve a confirmed complete response (CR) or partial response (PR), as assessed by investigators according to RECIST v1.1 criteria.

SECONDARY OUTCOMES:
Duration of Response (DoR) | From first documented response to progression or death (up to approximately 24 months)
  The time from the first documentation of CR or PR to the first documentation of disease progression or death from any cause, whichever occurs first, as assessed by investigators per RECIST v1.1.
Disease Control Rate (DCR) | From baseline to disease progression or end of treatment (up to approximately 24 months)
  The proportion of participants who achieve a best overall response of CR, PR, or stable disease (SD), as assessed by investigators using RECIST v1.1 criteria.
Progression-Free Survival (PFS) | From first dose until disease progression or death (up to approximately 24 months)
  Time from the date of first dose of study drug to the first documentation of disease progression or death from any cause, whichever occurs first, based on investigator assessment using RECIST v1.1.
Overall Survival (OS) | From first dose to death (up to approximately 36 months)
  Time from the date of first dose of study drug to death from any cause.
Frequency and Severity of Adverse Events (AEs) | From first dose through 30 days after the last dose of study treatment (up to approximately 30 months)
  Frequency and severity of treatment-emergent adverse events (TEAEs), treatment-related adverse events (TRAEs), serious adverse events (SAEs), and adverse events of special interest (AESIs), coded using MedDRA and graded per NCI-CTCAE v5.0.

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer center, Shanghai, China

IPD SHARING:
Plan to Share IPD: No